CLINICAL TRIAL: NCT03358251
Title: Investigation of the Safety and Efficacy of a Periodontal In-situ Gelling Product, Pocket-X Gel, in the Treatment of Periodontal Pockets Following Scaling and Root Planing
Brief Title: Investigation of the Safety and Efficacy of Pocket-X Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tree of Life Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PX-01
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SRP+Pocket-X Gel, split-mouth (Other): This arm is a split-mouth arm, i.e., participants will receive conventional treatment for periodontitis (scaling and root planing) for the entire mouth, and, in addition, will receive experimental treatment (Pocket-X Gel) for periodontal pockets present in one/two mouth segments (quadrants), while the contralateral quadrants will serve as control and will not undergo any further intervention.
  Interventions: Device: Pocket-X Gel; Procedure: Scaling and root planing

INTERVENTIONS:
Device: Pocket-X Gel — Pocket-X Gel is a biodegradable in-situ gelling product that is inserted into a pre-cleaned periodontal pocket where it quickly turns into a gel that adheres to the periodontal pocket and acts as a filler and physical barrier against bacterial re-colonization at the site of application. Administration of this product typically causes no discomfort. The product naturally degrades after 1-3 weeks.
Procedure: Scaling and root planing — Scaling and root planing is a conventional gold-standard treatment for periodontitis. As part of this procedure, subgingival plaque and tartar are removed and root surfaces are planed.

SUMMARY:
This study is an open-label split-mouth study in which Pocket-X Gel, a periodontal in-situ gelling product, will be applied to periodontal pockets in one/two mouth segment(s) of participants, following scaling and root planing on the entire mouth, while the contralateral segment(s) will serve as control. The aim of the study is to investigate the safety and efficacy of Pocket-X Gel in improving the healing of the gingiva and preventing bacterial re-colonization in the periodontal pocket following scaling and root planing.

DETAILED DESCRIPTION:
This study is an open-label split-mouth study that investigates the safety and efficacy of Pocket-X Gel, a periodontal in-situ gelling product, in improving the healing of the gingiva and preventing bacterial re-colonization in the periodontal pocket following scaling and root planing.

The study includes a single arm. All participants will undergo 1-4 sessions of scaling and root planing (SRP), which is the conventional gold-standard treatment for periodontal disease. The number of SRP sessions is dependent on the severity of the periodontal disease. Following completion of SRP, participants will undergo treatment with Pocket-X Gel, which will be inserted into periodontal pockets present in one/two of the participants mouth segments (quadrants), following scaling and root planing. The other mouth segments will not undergo further intervention. The number of segments to be treated is dependent on the clinical symmetry between the treated segment(s) and the contralateral segment(s). Participants will be followed for a total duration of 6 months. Additional application of Pocket-X Gel may occur 1 month and/or 3 months following first application, depending on the state of the participant's periodontal disease.

The rationale for the study is the hypothesis that a physical barrier inserted into periodontal pockets following scaling and root planing would assist in maintaining the pocket clean by preventing bacteria from re-entering the cleaned pocket, thus allowing the gums to properly heal and seal the pockets while preventing further inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Male or female, aged 18 and above
3. Provision of up-to-date full mouth periapical x-rays
4. Participants suffering from active moderate to severe chronic periodontitis with at least 3 sites of periodontal pockets of 5 mm or greater depth in each quadrant.
5. Participants with a minimum of 6 teeth with periodontal pocket depth of more than 5 mm.
6. Participants with a minimum of 20 teeth

Exclusion Criteria:

1. Known hypersensitivity to any of the devices components as listed on the user leaflet
2. Pregnancy or lactation
3. Smoking of more than 9 cigarettes per day
4. A concurrent dental disease, except for periodontitis, or planned treatment that may interfere with the study or study intervention, such as dental surgery, teeth implantation, etc.
5. Chronic disease such as diabetes mellitus or rheumatoid arthritis
6. Aggressive periodontitis
7. History of radiotherapy or chemotherapy
8. Immunodeficiency or autoimmune disease
9. Mental disorders
10. Parafunctional habits such as bruxism
11. Participant has taken antibiotics in the 6 months prior to the study
12. Participant has undergone periodontal treatment 12 months prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Hirsch, Principal Investigator — Dr. Ariel Hirsch Periodontal Clinic; Roni Kolerman, Principal Investigator — Dr. Roni Kolerman Periodontal Clinic
Locations (2):
- Israel (2):
  - Dr. Ariel Hirsch Periodontal Clinic, Tel Aviv
  - Dr. Roni Kolerman Periodontal Clinic, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Groups:
- SRP+Pocket-X Gel, Split-mouth: The single arm is a split-mouth arm, i.e., participants will receive conventional treatment for periodontitis (scaling and root planing) for the entire mouth, and, in addition, will receive experimental treatment (Pocket-X Gel) for periodontal pockets present in one/two mouth segments (quadrants), while the contralateral quadrants will serve as control and will not undergo any further intervention.
Period: Overall Study
Arm/Group | SRP+Pocket-X Gel, Split-mouth
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SRP+Pocket-X Gel, Split-mouth
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Periodontal Pockets Probing Depth
Description: Change in the probing depth of periodontal pockets which have undergone treatment with SRP+Pocket-X Gel in comparison to periodontal pockets which have undergone SRP only.
Time Frame: 12 and 24 weeks following first Pocket-X Gel administration
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: pockets
Groups:
- Lower Jaw Pockets + Treatment: Periodontal pockets situated in the lower jaw which received a treatment of SRP + Pocket-X gel.
- Lower Jaw Pockets - Control: Periodontal pockets situated in the lower jaw which received a tratment of SRP only.
- Upper Jaw Pockets + Treatment: Periodontal pockets situated in the upper jaw which received a treatment of SRP + Pocket-X gel.
- Upper Jaw Pockets + Control: Periodontal pockets situated in the upper jaw which received a treatment of SRP alone.
Arm/Group | Lower Jaw Pockets + Treatment | Lower Jaw Pockets - Control | Upper Jaw Pockets + Treatment | Upper Jaw Pockets + Control
Number analyzed (Participants) | 34 | 34 | 34 | 34
Number analyzed (pockets) | 63 | 63 | 109 | 109
mm
  depth at baseline | 6.97 (1.49) | 6.81 (1.59) | 7.67 (1.45) | 7.72 (1.30)
  depth at 3 months | 5.19 (0.98) | 5.69 (1.38) | 5.53 (1.07) | 6.35 (1.10)
  depth at 6 months | 4.5 (0.8) | 5.53 (1.24) | 4.74 (0.82) | 7.72 (0.99)

2. Secondary Outcome: Change in Clinical Attachment
Description: Change in the clinical attachment level of mouth segments which have undergone treatment with SRP+Pocket-X Gel in comparison to mouth segments which have undergone SRP only.
Time Frame: 12 and 24 weeks following first Pocket-X Gel administration
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: pockets
Arm/Group | Lower Jaw Pockets + Treatment | Lower Jaw Pockets - Control | Upper Jaw Pockets + Treatment | Upper Jaw Pockets + Control
Number analyzed (Participants) | 34 | 34 | 34 | 34
Number analyzed (pockets) | 63 | 63 | 109 | 109
mm
  change in CAL after 3 months | 2.08 (0.69) | 0.97 (0.64) | 2.62 (0.82) | 1.26 (0.68)
  change in CAL after 6 months | 3.01 (0.92) | 1.06 (0.63) | 3.61 (0.94) | 1.44 (0.83)

3. Secondary Outcome: Change in Recession Level
Description: Change in gingival recession level (buccal) of mouth segments which have undergone treatment with SRP+Pocket-X Gel in comparison to mouth segments which have undergone SRP only. Measured in mm.
Time Frame: 12 and 24 weeks following first Pocket-X Gel administration
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: pockets
Arm/Group | Lower Jaw Pockets + Treatment | Lower Jaw Pockets - Control | Upper Jaw Pockets + Treatment | Upper Jaw Pockets + Control
Number analyzed (Participants) | 34 | 34 | 34 | 34
Number analyzed (pockets) | 63 | 63 | 109 | 109
mm
  B recession at baseline | 1.36 (1.27) | 1.21 (1.17) | 1.49 (1.22) | 1.38 (1.06)
  B recession at 3 months | 1.06 (1.06) | 1.35 (1.32) | 1.01 (0.98) | 1.49 (1.24)
  B recession at 6 months | 0.82 (0.89) | 1.43 (1.42) | 0.80 (0.88) | 1.51 (1.38)

4. Secondary Outcome: Change in Bleeding Index
Description: Change in gingival bleeding index of mouth segments which have undergone treatment with SRP+Pocket-X Gel in comparison to mouth segments which have undergone SRP only.
Time Frame: 12 and 24 weeks following first Pocket-X Gel administration
Measure: Number; unit: % percent of pockets bleeding
Units Other Than Participants: pockets
Arm/Group | Lower Jaw Pockets + Treatment | Lower Jaw Pockets - Control | Upper Jaw Pockets + Treatment | Upper Jaw Pockets + Control
Number analyzed (Participants) | 34 | 34 | 34 | 34
Number analyzed (pockets) | 63 | 63 | 109 | 109
% percent of pockets bleeding
  percent of pockets bleeding at baseline | 98.4 | 85.7 | 92.66 | 92.66
  percent of pockets bleeding after 3 months | 20.63 | 36.51 | 20.18 | 45.87
  percent of pockets bleeding after 6 months | 12.70 | 28.57 | 8.33 | 44.44

5. Secondary Outcome: Change in Mobility Grade
Description: Change in mobility grade of teeth present in mouth segments which have undergone treatment with SRP+Pocket-X Gel in comparison to mouth segments which have undergone SRP only.
  Mobility is graded clinically by applying pressure with the ends of 2 metal instruments (e.g. dental mirrors) and trying to rock a tooth gently in a bucco-lingual direction (towards the tongue and outwards again).
  Normal, physiologic tooth mobility of about 0.25 mm is present in health. This is because the tooth is not fused to the bones of the jaws, but is connected to the sockets by the periodontal ligament.
  Abnormal, pathologic tooth mobility occurs when the attachment of the periodontal ligament to the tooth is reduced (attachment loss), or if the periodontal ligament is inflamed. Tooth mobility is measured and graduated from 0-3.
  Grade 0: No apparent mobility Grade 1: Perceptible mobility <1mm in buccolingual direction Grade 2: >1mm but <2mm Grade 3: >2mm or depressibility in the socket
Time Frame: 12 and 24 weeks following first Pocket-X Gel administration
Measure: Mean (Standard Deviation); unit: mobility grade
Units Other Than Participants: pockets
Arm/Group | Lower Jaw Pockets + Treatment | Lower Jaw Pockets - Control | Upper Jaw Pockets + Treatment | Upper Jaw Pockets + Control
Number analyzed (Participants) | 34 | 34 | 34 | 34
Number analyzed (pockets) | 63 | 63 | 109 | 109
mobility grade
  Mobility at baseline | 0.19 (0.50) | 0.19 (0.53) | 0.18 (0.51) | 0.19 (0.52)
  Mobility after 3 months | 0.05 (0.21) | 0.14 (0.50) | 0.05 (0.23) | 0.15 (0.38)
  Mobility after 6 months | 0 (0) | 0.01 (0.12) | 0.01 (0.10) | 0.12 (0.35)

ADVERSE EVENTS:
Time Frame: until the last visit of the patient, 6 month post the first application of the treatment.
Arm/Group | SRP+Pocket-X Gel, Split-mouth
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT03358251/Prot_SAP_000.pdf